CLINICAL TRIAL: NCT01133106
Title: Psychosocial/Behavioral Intervention in Post-Stroke Depression (PSD)
Brief Title: Living Well With Stroke
Acronym: PSD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Pamela Mitchell, Professor, School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37952-J; R01NR007755 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Cerebrovascular Stroke; Depression
Keywords: stroke recovery; quality of life
MeSH Terms: conditions — Stroke; Depression | interventions — Behavior Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- In-person behavioral intervention (Experimental): behavioral counseling plus antidepressant treatment prescribed by participant's own provider; consisted of orientation session plus 6 counseling sessions in person with a psychosocial nurse practitioner
  Interventions: Behavioral: Brief pleasurable events/behavioral therapy
- Telephone behavioral intervention (Experimental): This arm is identical to the in-person Arm except that the intervention is delivered by telephone instead of in-person.
  Interventions: Behavioral: Brief pleasurable events/behavioral therapy
- Standard care (Active Comparator): participants have orientation to the study with the same written materials given those in the experimental arms. Keep a medication log and keep appointments with their own post-stroke provider
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: Brief pleasurable events/behavioral therapy — Each participant in any arm will be given an American Stroke Association article about stroke and depression, a Stroke Smart Article about caregiver depression, and a pamphlet by the Beck Institute titled "Coping with Depression".
  Each participant in Arms 1 and 2 will be given their own manual for the intervention sessions. The intervention consists of one in-person orientation session and 6 weekly sessions with the following topics introducing behavioral therapy, the role of pleasant events, problem-solving skills and generalization techniques. All participants' primary care provider or stroke care provider will receive a letter informing them of their patient's participation (but not of study assignment). This letter will include recommendations for prescribing and adjusting antidepressant treatment using established guidelines adapted for treatment of medically-ill outpatients.
  Arms: In-person behavioral intervention; Telephone behavioral intervention
Other: Standard care — The standard care group (Arm C, N=75) will receive standard medical treatment from their provider, including a recommendation for antidepressants. Participants or third-party payers will pay for their antidepressants, just as they would under regular care. All participants receive written materials regarding depression from the American Stroke Association, keep medication logs and receive follow-up assessment on the same time frame as the intervention groups
  Arms: Standard care

SUMMARY:
The overall goal of this study is to conduct a three-armed randomized controlled trial (RCT) in stroke survivors with depression to determine if a brief psychosocial-behavioral therapy intervention delivered in-person (arm A) or by telephone (arm B) is better than usual care (arm C), in terms of percent reduction in depressive symptoms and % of participants achieving remission of symptoms.

DETAILED DESCRIPTION:
This is the second phase of a study whose aim was to evaluate the short and long-term efficacy of a brief psychosocial/behavioral intervention (with adjunctive antidepressant)for the treatment of post-stroke depression (PSD) in survivors of ischemic stroke (registered as clinical trail NCT00194454). In the earlier trial we demonstrated that a pleasant event/problem-solving brief psychosocial-behavioral therapy delivered by psychosocial nurse practitioners was highly effective in treating major depression and promoting remission in ischemic stroke survivors for up to two years. In this phase, we refine the protocol, and potentially make it more cost effective, by conducting a randomized comparative effectiveness trial of in-person versus telephone delivery of the intervention, comparing with usual care control. We also seek to expand our sample to include hemorrhagic stroke survivors (intraparenchymal hemorrhage and subarachnoid hemorrhage) as well as those with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for an ischemic or hemorrhagic stroke (intraparenchymal hemorrhage- IPH or subarachnoid hemorrhage - SAH) in the past 3 months
* clinical depression symptoms (Geriatric Depression Score -GDS >= 11

Exclusion Criteria:

* major psychiatric co-morbidity
* active suicidal ideation without ability to contract for safety
* current substance abuse
* physical inability to tolerate 1-2 hour sessions
* receptive or global aphasia
* reduced level of consciousness (GCS<15).

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD) | 1 year post-treatment
  Remission is defined as an HRSD score of 9 or less on the 17 item scale

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | 1 year post treatment
  The SIS has multiple scales measuring limitations in activity, in social participation and perceived overall stroke impact (perceived percent recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela H Mitchell, PhD, Principal Investigator — University of Washington; Catherine J Kirkness, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be provided to qualified investigators, including students conducting secondary analysis

REFERENCES:
- [Background] Mitchell PH, Veith RC, Becker KJ, Buzaitis A, Cain KC, Fruin M, Tirschwell D, Teri L. Brief psychosocial-behavioral intervention with antidepressant reduces poststroke depression significantly more than usual care with antidepressant: living well with stroke: randomized, controlled trial. Stroke. 2009 Sep;40(9):3073-8. doi: 10.1161/STROKEAHA.109.549808. Epub 2009 Aug 6. PMID 19661478
- [Background] Mitchell PH, Teri L, Veith R, Buzaitis A, Tirschwell D, Becker K, Fruin M, Kohen R, Cain KC. Living well with stroke: design and methods for a randomized controlled trial of a psychosocial behavioral intervention for poststroke depression. J Stroke Cerebrovasc Dis. 2008 May-Jun;17(3):109-15. doi: 10.1016/j.jstrokecerebrovasdis.2007.12.002. PMID 18436150
- [Result] Kirkness, CJ, Buzaitis, A, Habermann, B, Jessup, NM, McClennon, SM, McKenzie, S, Weaver, M, Weisman, P, Mitchell PH, Bakas, T. (2014) Methodological issues in telephone interventions for stroke survivors and family caregivers. Abstract 86. Stroke. 45(Suppl_1) (Supplement 1):A86, February 2014
- [Result] Kirkness CJ, Becker KJ, Cain KC, Kohen, R, Tirschwell, DL, Teri L, Veith RR, Mitchell PH (2015) Telephone versus in-person psychosocial behavioral treatment in post-stroke depression. Abstract WP:125. Stroke 46 (supplement 1): WP 125, February 2015. http://stroke.ahajournals.org/content/46/Suppl_1/AWP125.abstract?sid=441a6914-e14e-4969-85f9-964367d56ed7
- [Derived] Byun E, Becker KJ, Kohen R, Kirkness CJ, Mitchell PH. Brief Psychosocial Intervention to Address Poststroke Depression May Also Benefit Fatigue and Sleep-Wake Disturbance. Rehabil Nurs. 2021 Jul-Aug 01;46(4):222-231. doi: 10.1097/RNJ.0000000000000304. PMID 33443981
- [Derived] Byun E, Kohen R, Becker KJ, Kirkness CJ, Khot S, Mitchell PH. Stroke impact symptoms are associated with sleep-related impairment. Heart Lung. 2020 Mar-Apr;49(2):117-122. doi: 10.1016/j.hrtlng.2019.10.010. Epub 2019 Dec 12. PMID 31839325
- [Derived] Kirkness CJ, Cain KC, Becker KJ, Tirschwell DL, Buzaitis AM, Weisman PL, McKenzie S, Teri L, Kohen R, Veith RC, Mitchell PH. Randomized trial of telephone versus in-person delivery of a brief psychosocial intervention in post-stroke depression. BMC Res Notes. 2017 Oct 10;10(1):500. doi: 10.1186/s13104-017-2819-y. PMID 29017589